CLINICAL TRIAL: NCT07375420
Title: Optimising Prehabilitation Exercise to Enhance Tumour Outcomes in Advanced Oesophageal Cancer
Brief Title: Will a Pre-therapy Exercise Intervention Improve the Outcomes of Patients With Advanced Oesophageal Cancer?
Acronym: OPTIMUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Collaborators: World Cancer Research Fund International (Other)
Responsible Party: Principal Investigator, Adam Frampton, Professor Adam Frampton, University of Surrey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 326527
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Oesophageal Adenocarcinoma; T Cells; Tumor Microenvironment; Exercise
Keywords: oesophageal cancer; exercise; tumour microenvironment
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Motor Activity; Esophageal Neoplasms | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low intensity/Low amount (LAM) arm (Active Comparator)
  Interventions: Behavioral: Low intensity exercise
- moderate-vigorous-intensity/moderate-high-amount (MAM) arm (Experimental)
  Interventions: Behavioral: High intensity exercise

INTERVENTIONS:
Behavioral: Low intensity exercise — Participants undertake supervised cycling twice weekly. Each session comprises 5 min warm-up at 30% heart rate reserve (HRR), then 20 min continuous cycling starting at 40% HRR. After participants complete two supervised sessions/week at 40% HRR without adverse events, intensity increases by 5% HRR per session to a target of 60% HRR, which is maintained for the remainder of the pre-operative period (until surgery). After cycling, participants complete flexibility and resistance exercises targeting six major muscle groups (2 sets of 12 repetitions, rating of perceived exertion (RPE) 12-14), with load increased when RPE <12. Participants also complete a home programme three times weekly (60 min/session) focusing on resistance and core stability using appropriately weighted bands.
  Arms: Low intensity/Low amount (LAM) arm
Behavioral: High intensity exercise — Exercise Group 2 (moderate-vigorous-intensity/moderate-high-amount (MAM)) is a progressive, individualised programme with two supervised aerobic sessions/week using harness-supported treadmill walking where possible, or cycle ergometry if needed. Each session begins with 5 min at 40% heart rate reserve (HRR). For ~2 weeks, participants complete 15 min of intervals (30 s at 80% HRR then 1 min at 50% HRR), followed by 5 min cool-down at 40% HRR. Training then progresses by increasing hard bouts to 1 min, building to 20 intervals, then targeting 90%/50% HRR with gradual increases in time spent at 90% HRR. After aerobic exercise, flexibility plus resistance (chest press, leg press, seated row) is performed for 2 sets to fatigue at rating of perceived exertion (RPE) 15-17, increasing load when 2x25 reps are achieved. Home aerobic exercise is prescribed for 60 min, 3x/week at ~60% HRR using heart-rate telemetry (home cycle provided if walking not feasible).
  Arms: moderate-vigorous-intensity/moderate-high-amount (MAM) arm

SUMMARY:
Background

Regular exercise can significantly improve physical and mental health during cancer treatment and reduce the time needed in the hospital. Animal studies suggest that exercise training can also reduce the number of cancer cells. For example, exercise training in mice produces more immune cells in the tumour. These immune cells in the tumour contribute to the destruction and reduction of the size of the tumour and are a vital component of effective immunotherapy (cancer treatment that helps the immune system fight cancer).

In humans, exercise training and the immune response in tumours are less understood. Only 1 study has investigated the effect of a single exercise session before surgical removal of the prostate in prostate cancer patients. As the benefits of exercise are gained from weeks/months of exercise, no effect on the immune cells in the tumours were found.

The investigators have carried out a previous study looking at how exercise affects fitness before major surgery. After this they used state-of-the-art methods to detect and visualise immune cells within the tumour. Compared with the patients who did not exercise, the exercise group had significantly more immune cells in their tumours, consisting of a group of cells that are important for killing cancerous cells called CD8+ T cells. CD8+ T cells in tumours are associated with improved survival outcomes.

Importantly, they found a link between changes in fitness and the amount of these cells in the tumour. This suggests that if there is increase in fitness, there also an increase in the frequency of these cells in the tumour. Therefore, the investigators propose performing a clinical trial to find out the best level of exercise patients need to sustain before surgery to produce this improved immune response.

The trial will aim to understand how this happens and how the entry of immune cells into the tumour changes the environment around a tumour. The investigators consist of a team of exercise immunologists, tumour immunologists and clinicians working with the Human Performance Institute at the University of Surrey in collaboration with the Royal Surrey NHS Trust.

How it will be done

The investigators will assess immune cell response in blood samples obtained from oesophageal cancer patients before, during and after a high or low intensity exercise programme. Following the exercise programme, tumour tissue removed at surgery from these patients will be used to investigate the the presence and quantity of these immune cells.

Potential impact

A better understanding of this is important, as current anti-cancer immune-based therapeutics work best when there is a an immune response within the patient's tumour. Generating evidence that exercise can improve the immune response against the tumour in patients with oesophageal cancer would provide significant justification for introducing "personalised" exercise programmes to improve treatment outcomes.

DETAILED DESCRIPTION:
Oesophageal cancer is one of the most challenging cancers to treat, with low survival rates, even when people receive intensive treatments such as chemotherapy and surgery. New treatment strategies could therefore lead to significant benefits to patients.

One of the most promising new treatments is immunotherapy, which works by "releasing the brakes" on immune cells. Immunotherapy has transformed outcomes in some cancers, but its impact in oesophageal cancer has been modest so far. One important reason may be that many oesophageal tumours contain few active immune cells to begin with. Finding safe, practical ways to ''wake up'' the immune system and draw immune cells into the tumour could make existing treatments more effective.

Exercise is a simple, low-cost option that could help. Exercise programmes are already used before major surgery to improve fitness and help people cope better with treatment. Research in other cancers shows that exercise can increase the number and activity of key immune cells in the blood and, in some cases, inside tumours. Exercise also affects the gut microbiome. This is the community of bacteria and other microorganisms in our intestines, and the chemicals they produce. These microbial products can travel through the bloodstream and shape how the immune system behaves. However, it is still unclear yhow these changes work together in people with oesophageal cancer receiving chemotherapy.

In this study, people with oesophageal cancer who are due to receive chemotherapy before surgery will be invited to join a supervised exercise programme. All patients will exercise under the guidance of specialist staff while they are on chemotherapy. One group will follow a lower-intensity programme similar to current NHS prehabilitation. The other group will complete higher-intensity sessions, within safe limits. Comparing these two realistic options will allow us to test whether exercise intensity makes a difference.

The investigators will collect blood and stool samples at key time points before and during treatment. From blood, there will be an analysis of the changes in immune cells and proteins that signal how "switched on" the immune system is. From stool, the investigators will study the gut microbiome and the metabolites (small molecules) they produce. After surgery, the removed tumour will be examined under the microscope to see whether exercise is linked to differences in the number and type of immune cells inside the tumour. By bringing these measurements together, we hope to understand whether more intensive exercise leads to a more immune-active tumour, and how the change in immune cells alongside systemic signalling molecules are related to these states.

ELIGIBILITY:
Inclusion Criteria:

* Adults with resectable oesophageal adenocarcinoma who are planned for neoadjuvant chemotherapy followed by surgery

Exclusion Criteria:

* Inability to carry out CPET or exercise due to underlying health conditions
* pregnancy
* <18 years old

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-26 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Tumour immune infiltration | From enrollment to the end of treatment at 16 weeks
  Percentage increase of CD8 T Cells within the tumour
Improvement in cardiorespiratory function | From enrollment to the end of treatment at 16 weeks
  Measured through VO2 peak

SECONDARY OUTCOMES:
Change in peripheral blood mononuclear cells (PBMC) | From enrollment to the end of treatment at 16 weeks
  We will analyse longitudinal shifts in PBMC subsets and phenotypes.
Change in plasma cytokines | From enrollment to the end of treatment at 16 weeks
  We will analyse longitudinal shifts in PBMC subsets and phenotypes.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Frampton, PhD, Principal Investigator — University of Surrey
Locations (1):
- University of Surrey, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes